CLINICAL TRIAL: NCT00236964
Title: Comparison of Oral Iron With IV Iron in Patients With Anemia of Chronic Renal Failure Not on Dialysis
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: American Regent, Inc. (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 1VEN99012
Record Dates: First submitted 2005-10-07; First posted 2005-10-12 (Estimated); Last update posted 2025-05-09 (Actual); Status verified 2018-01

CONDITIONS: Anemia
Keywords: Anemia; Chronic Kidney Disease
MeSH Terms: conditions — Anemia; Renal Insufficiency, Chronic | interventions — Ferric Oxide, Saccharated; Erythropoietin; Iron; ferrous sulfate

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- Iron Sucrose (Experimental): Iron sucrose 200 mg intravenous on Days 1, 8, 15, 22, and 29
  Interventions: Drug: Iron Sucrose + Erythropoietin
- Oral Iron (Active Comparator): Oral ferrous sulfate 325 mg three times a day on Days 1 to 29.
  Interventions: Drug: Oral Iron + Erythropoietin

INTERVENTIONS:
Drug: Iron Sucrose + Erythropoietin — The total dose of iron sucrose was 1,000 mg. Participants also received erythropoietin 2,000 units subcutaneously on Days 1, 8, 15, 22, 29, and 36.
  Other Names: Venofer
  Arms: Iron Sucrose
Drug: Oral Iron + Erythropoietin — Oral iron 325 mg three time daily for 29 days. Participants also received erythropoietin 2,000 units subcutaneously on Days 1, 8, 15, 22, 29, and 36.
  Other Names: Ferrous sulfate
  Arms: Oral Iron

SUMMARY:
The purpose of the study was to compare the efficacy of oral iron (ferrous sulfate) plus erythropoietin to Iron Sucrose plus erythropoietin for managing anemia patients with chronic renal failure who are not receiving dialysis.

DETAILED DESCRIPTION:
Randomized open-label multicenter active-controlled study of anemic patients with Chronic Renal Failure who are not yet receiving dialysis. The duration of the study was five months. After screening procedures including multiple hemoglobin values, patients were randomly assigned to either IV Iron Sucrose (200mg X 5) or oral iron sulfate (325mg TID)for 29 days. Safety assessments included the recording of all adverse events, physical examinations, vital signs, electrocardiograms and clinical laboratory tests. Efficacy parameters included hematologic parameters.

ELIGIBILITY:
Inclusion Criteria:

* Creatine Clearance <40 mL/min
* Average Baseline Hemoglobin < 10.5g/dL
* Serum Transferrin Saturation (TSAT) < 25% and Ferritin <300ng/mL

Exclusion Criteria:

* Blood Transfusion within 30days
* Uncontrolled Hypertension
* Suffering form concommitant disease of the liver
* Serious bacterial infection
* Pregnancy / lactation
* Symptomatic HIV
* Expected to under dialysis or renal transplant during study

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 96 (Actual)
Dates: Start 2001-02-23 (Actual); Primary Completion 2002-05-30 (Actual); Study Completion 2002-05-30 (Actual)

PRIMARY OUTCOMES:
Mean Change in Hemoglobin | Baseline and Day 43
  Change in hemoglobin g/dL from baseline to Day 43 was analyzed using parametric analysis of covariance (ANCOVA).
Mean Change in Serum Ferritin | Baseline and Day 43
  Change in Ferritin ng/mL from baseline to Day 43 was analyzed using parametric analysis of covariance (ANCOVA).

SECONDARY OUTCOMES:
Clinical Success (Change in Hemoglobin) | Baseline and Day 43
  Participants were considered to have achieved clinical success if they attained a change in hemoglobin ≥0.8 g/dL. The difference from baseline to Day 43 was calculated and rounded.
Clinical success (change in Ferritin) | Baseline and Day 43
  Participants were considered to have achieved clinical success if they attained a change in ferritin ≥160 ng/mL. The difference from baseline to Day 43 was calculated and rounded.

CONTACTS AND LOCATIONS:
Overall Officials: Mark Falone, MD, Study Director — Medical Director

REFERENCES:
- [Result] Charytan C, Qunibi W, Bailie GR; Venofer Clinical Studies Group. Comparison of intravenous iron sucrose to oral iron in the treatment of anemic patients with chronic kidney disease not on dialysis. Nephron Clin Pract. 2005;100(3):c55-62. doi: 10.1159/000085049. Epub 2005 Apr 11. PMID 15824508